CLINICAL TRIAL: NCT01555905
Title: Respiratory Muscle Strength and Function in Patients With Neuromuscular Disease
Brief Title: Respiratory Muscle Strength in Patients With NMD
Acronym: RMST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB201600270
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Neuromuscular Disease
Keywords: Respiratory Muscle Strength
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Exercise (Experimental): Threshold PEP or IMT device Phillips-Respironics
  Interventions: Device: Threshold PEP or IMT device Phillips-Respironics

INTERVENTIONS:
Device: Threshold PEP or IMT device Phillips-Respironics — The subject will be instructed to take 8-15 deep, forceful breaths through the Threshold device, followed by at least 3 minutes of rest. The process will be repeated 3 more times for a total of 4 sets of 8-15 breaths. IMST will be completed three to five days per week, based upon the subject's daily baseline level of fatigue.

SUMMARY:
The purpose of this study is to determine if inspiratory muscle strength training (IMST) will impact maximal inspiratory pressure and pulmonary function in patients with neuromuscular disease.

DETAILED DESCRIPTION:
Subjects undergo a 12-week period of inspiratory muscle strength training. Respiratory strength is assessed before and after the training period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of neuromuscular disease
* Clinical evidence of impaired pulmonary function

Exclusion Criteria:

* Above or below age range
* No clinical evidence of impaired pulmonary function
* No diagnosis of a neuromusuclar disease
* Presence of an acute illness at time of study
* Participating in other research studies involving investigational drugs
* Diagnosis of a primary pulmonary disease
* Use of tobacco products

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Smith, PhD, PT, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise
Started | 17
Completed | 7
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Exercise
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 24 [1 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Maximal Inspiratory Pressure [Mean (Full Range); unit: cm H2O] | 37.3 [9.8 to 71]

OUTCOME MEASURES:

1. Primary Outcome: Maximal Inspiratory Pressure
Description: The primary endpoints for inspiratory muscle training efficacy will be maximal inspiratory pressure tests, a measure of respiratory strength.
Time Frame: Baseline (pre-IMST) and 3 months (post-IMST)
Measure: Mean (Full Range); unit: cm H2O
Arm/Group | Exercise
Number analyzed (Participants) | 7
cm H2O
  Pre | 33.7 [9.8 to 68]
  Post | 38.0 [12.8 to 65]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Exercise
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise (N=17)
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study termination due to low proportion of subjects who completed the intervention and returned to the study center for post-testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT01555905/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT01555905/ICF_001.pdf